CLINICAL TRIAL: NCT04374864
Title: Dose of Trelagliptin for Egyptian Patients Requires no Modification Than Japanese
Brief Title: Dose Modification Requirement for Trelagliptin in Egyptian Population
Acronym: Trelagliptin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: British University In Egypt (Other)
Collaborators: Nermeen Ashoush (Unknown); Shereen Mowaka (Unknown); Mariam M. Tadros (Unknown)
Responsible Party: Principal Investigator, Bassam Mahfouz Ayoub, Associate Professor in Pharmaceutical Department, British University In Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BUE 2020
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — trelagliptin

STUDY DESIGN:
Intervention Model Description: Good health of the human subjects was confirmed with a complete medical history and physical examination. Fasting of all volunteers eliminated the possible interaction from high fat meals. The evaluation of safety of the study was based on monitoring of blood glucose level, vital signs, pulse rate, monitoring of adverse events, and physical examination. Samples from 6 healthy, adult, male, Egyptian volunteers (age: 25-39 years, average weight: 89.8 kg, average body mass index (BMI): 34.2) were collected at 0, 0.5, 1, 1.5, 2, 2.5, 3, 8, 24, 48, 72, 96, 120, 144 and 168 hrs, transferred to heparinized centrifuge tubes and analyzed with the proposed method after single oral dose administration of one Zafatek® tablet nominally containing 50 mg TLN. Blood samples (1 mL of each sample) were centrifuged at 3000 rpm for 5 min.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trilaglibtin 50 mg (Experimental): Samples from 6 healthy, adult, male, Egyptian volunteers (age: 25-39 years, average weight: 89.8 kg, average body mass index (BMI): 34.2) were collected at 0, 0.5, 1, 1.5, 2, 2.5, 3, 8, 24, 48, 72, 96, 120, 144 and 168 hrs, transferred to heparinized centrifuge tubes and analyzed with the proposed method after single oral dose administration of one Zafatek® tablet nominally containing 50 mg trilagliptin. Blood samples (1 mL of each sample) were centrifuged at 3000 rpm for 5 min.
  Interventions: Drug: Trelagliptin

INTERVENTIONS:
Drug: Trelagliptin — Anti diabetic

SUMMARY:
The proposed study will consider the pharmacokinetic evaluation of Trelagliptin after administration to Egyptian volunteers and the results will be compared with the other reported ethnic populations. The FDA recognizes that standard methods of defining racial subgroups are necessary to compare results across pharmacokinetic studies, and to assess potential subgroup differences. The design of the study is open labeled, one treatment, one period, single dose pharmacokinetic study.

DETAILED DESCRIPTION:
The proposed study will consider the pharmacokinetic evaluation of Trelagliptin after administration to Egyptian volunteers and the results will be compared with the other reported ethnic populations. The FDA recognizes that standard methods of defining racial subgroups are necessary to compare results across pharmacokinetic studies, and to assess potential subgroup differences. The design of the study is open labeled, one treatment, one period, single dose pharmacokinetic study. The main pharmacokinetic parameters which are Cmax, Tmax, t1/2, elimination rate constant, AUC0-t and AUC0-inf, will be estimated. Fasting of all volunteers will eliminate the possible interaction from food or caffeine consumption. The pharmacokinetic parameters of Trelagliptin will be studied in healthy human subjects according to the ethical regulations of World Medical Association Declaration of Helsinki (October 1996) and the International Conference of Harmonisation Tripartite Guideline for Good Clinical Practice. Written informed consent was provided (attached and signed by the six volunteers) in order to be approved by the ethics committee of the Faculty of Pharmacy, The British University in Egypt. The good health of the human subjects was confirmed by a complete medical history and physical examination. Samples from six, healthy, adult, male, smoking, Egyptian volunteers (age: 25-39 years, average weight: 89.8 kg, Average BMI: 34.2) will be collected at 0, 0.5, 1, 1.5, 2, 2.5, 3, 8, 24, 48, 72, 96, 120, 144 and 168 hrs to be transferred to heparinized centrifuge tubes in order to be analyzed by LC-MS/MS study (developed & validated) after single oral dose administration of one Zafatek® tablet nominally containing 50 mg Trelaglipitin. The blood samples (1 mL of each sample) will be centrifuged at 3000 rpm for 5 minutes, The main pharmacokinetic parameters of the study which are Cmax, Tmax, t1/2, elimination rate constant, AUC0-t and AUC0-inf will be estimated, using a validated excel software. Blood glucose level will be determined for all volunteers at different time intervals to monitor any hypoglycemic effect. The study will be conducted as per FDA guidelines. The development of such correlations between trelagliptin concentrations and its pharmacologic responses will enable clinicians to apply pharmacokinetic principles to actual patient situations. The evaluation of safety of the study will be based on monitoring of blood glucose level, vital signs, pulse rate, monitoring of adverse events, and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* The good health of the human subjects was confirmed by a complete medical history and physical examination.

Exclusion Criteria:

* Patients suffering from any chronic disease other than diabetes will be excluded from the study.

Ages: 25 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Cmax | 12 hours
  The peak plasma concentration of a drug after administration
Tmax | 12 hours
  Time to reach Cmax.
Elimination half life | 12 hours
  The time required for the concentration of the drug to reach half of its original value.
Elimination rate constant | 12 hours
  The rate at which a drug is removed from the body.
Area under the curve | 12 hours
  The integral of the concentration-time curve

CONTACTS AND LOCATIONS:
Locations (1):
- The British University in Egypt, Cairo, El Sherouk, Egypt

IPD SHARING:
Plan to Share IPD: Undecided